CLINICAL TRIAL: NCT06354244
Title: Effects of Electroacupuncture of Different Treatment Frequency in Chronic Urinary Retention Caused by Lower Motor Neuron Lesions: a Prospective Cohort Study
Brief Title: Electroacupuncture of Different Treatment Frequency in Chronic Urinary Retention Caused by Lower Motor Neuron Lesions
Status: Recruiting | Type: Observational
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 2023-183-KY-02
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Urinary Retention; Lower Motor Neurone Lesion
Keywords: electroacupuncture; chronic urinary retention; cohort study
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Electroacupuncture of 2 sessions per week
  Interventions: Device: Electroacupuncture of 2 sessions per week
- Electroacupuncture of 3 sessions per week
  Interventions: Device: Electroacupuncture of 3 sessions per week
- Electroacupuncture of 4 sessions per week
  Interventions: Device: Electroacupuncture of 4 sessions per week

INTERVENTIONS:
Device: Electroacupuncture of 2 sessions per week — Acupoints including bilateral BL23, BL32, BL33, BL35 and SP6 are inserted with acupuncture needles(size 0.30 × 40 mm and 0.30 × 75 mm or 0.40 × 100 mm,Hwato Brand). Bilateral BL32 and BL33 are needled to a depth of 70-95 mm with an angle of 60°-75° inward and downward, into the second and third sacral foramen. Bilateral BL35 are needled to a depth of 60-70 mm in a slightly superolateral direction. Bilateral BL23 and SP6 are vertically needled to a depth of 25-30 mm. After deqi is evoked, electric stimulators with a 5Hz continuous wave (5-10 mA intensity) are separately connected to bilateral BL32, BL33,BL35 and SP6. Current intensity is adjusted according to the patients' individual tolerance. During each session, electroacupuncture(EA) is retained for 30 minutes. The patients receive EA 2 sessions per week for 2-24 weeks.EA can be terminated if the patient acquire satisfactory spontaneous urination.
  Groups: Electroacupuncture of 2 sessions per week
Device: Electroacupuncture of 3 sessions per week — Acupoints and electroacupuncture (EA) procedures are the same as in the group of EA of 2 sessions per week, but the patients receive EA 3 sessions per week for 2-24 weeks in this group.EA can be terminated if the patient acquire satisfactory spontaneous urination.
  Groups: Electroacupuncture of 3 sessions per week
Device: Electroacupuncture of 4 sessions per week — Acupoints and electroacupuncture (EA) procedures are the same as in the group of EA of 2 sessions per week, but the patients receive EA 4 sessions per week for 2-24 weeks in this group.EA can be terminated if the patient acquire satisfactory spontaneous urination.
  Groups: Electroacupuncture of 4 sessions per week

SUMMARY:
The aim of this study is to compare the effects of electroacupuncture of different frequency in patients with chronic urinary retention caused by lower motor neuron lesions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with urinary retention caused by lower motor neuron lesions (e.g., sacral plexus, cauda equina, or sacral cord lesions).
* 18 years or older.
* Baseline post void residuals (PVR) ≥150 mL.
* The course of urinary retention ≥1 month.
* Having normal bladder sensation.
* Using clean intermittent catheterization (CIC), indwelling catheterization (IC), manual assisted voiding including putting pressure on abdomen, or cystostomy catheterization.
* Signed informed consent and voluntary participation in the study.

Exclusion Criteria:

* Having a lower urinary tract obstruction, such as bladder neck contracture, urethral stricture, prostatic hyperplasia, or large urinary stones that can cause obstruction.
* Having any type of malignant tumors not removed.
* Having severe systemic disorders not controlled.
* Having implanted electrodes of cardiac pacemaker, pudendal nerve stimulation, bladder stimulation, or SNM.
* Pregnancy or lactation.
* Eletroacupuncture treatment duration < 2 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are a group of patients with nerve lesions presenting with chronic urinary retention, having to rely on life-long catheterization to empty the bladder. However, complications of catheterization including recurrent urinary tract infection and urethral stricture formation, negatively impact on patients' daily life and bring heavy burden on family and society, together making it a less ideal option.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The response rate. | Week 12.
  Responders are defined as patients whose post void residuals (PVR) reduced by 50% or more from baseline.

SECONDARY OUTCOMES:
The response rate. | Week 4, Week 8 and Week 24.
  Responders are defined as patients whose post void residuals (PVR) reduced by 50% or more from baseline.
The change in post void residuals (PVR) from baseline. | Week 4, Week 8,Week 12 and Week 24.
  PVR is measured by urethral catheter output after patients' spontaneous urination attempts without catheterization or assisted bladder emptying (including increasing abdominal pressure or other auxiliary manual methods). If catheterization is not needed, which is assessed by urologists, PVR will be measured by ultrasound.
The change in the proportion of patients reporting severe urinating difficulty from baseline. | Week 4, Week 8,Week 12 and Week 24.
  The patient' s urinating difficulty is classified into four levels: severe, moderate, mild and none.
The change in the proportion of patients having stool retention from baseline. | Week 4, Week 8,Week 12 and Week 24.
  Stool retention is diagnosed according to Rome IV criteria.
The change in the proportion of patients requiring catheterization from baseline. | Week 4, Week 8,Week 12 and Week 24.
  If satisfactory spontaneous urination is observed,catheterization will not be needed, which is assessed by urologists.
The proportion of patients reporting much better or moderately better regarding the Patient Global Impression of Improvement (PGI-I). | Week 4, Week 8,Week 12 and Week 24.
  The PGI-I assessment has scores of 1 to 7 corresponding to much better to much worse, with higher score representing less improvement.
The proportion of patients having recurrent symptomatic UTI, hydroureter, or hydronephrosis. | Week 4, Week 8,Week 12 and Week 24.
  Recurrent UTI is confirmed by characteristic clinical signs.Hydronephrosis and hydroureter are assessed by ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with the publication until six months after publication.
  A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal.
  Researchers whose proposal has been approved will sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with the publication until six months after publication.
Access Criteria: A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal. Researchers whose proposal has been approved.
  Researchers whose proposal has been approved will sign a data access agreement.